CLINICAL TRIAL: NCT03523260
Title: High-Flow Hemodialysis Catheters Placed Through the Left Internal Jugular Approach (R12-022)
Brief Title: Comparison of High-Flow Hemodialysis Catheters Placed From the Left Internal Jugular Vein(R12-022)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never funded
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Husameddin M El Khudari, Interventional Radiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-130430002
Record Dates: First submitted 2018-02-07; First posted 2018-05-14 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: End Stage Renal Disease on Dialysis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Tunneled dialysis Split-tip catheter (Active Comparator): High-flow tunneled Split-tip catheter for hemodialysis will be inserted by standard interventional technique
  Interventions: Device: Tunneled dialysis catheter placement.
- Tunneled dialysis Step-tip catheter (Active Comparator): High-flow tunneled Step-tip catheter for hemodialysis will be inserted by standard interventional technique
  Interventions: Device: Tunneled dialysis catheter placement.
- Tunneled dialysis Symmetric tip catheter (Active Comparator): High-flow tunneled Symmetric tip catheter for hemodialysis will be inserted by standard interventional technique
  Interventions: Device: Tunneled dialysis catheter placement.

INTERVENTIONS:
Device: Tunneled dialysis catheter placement. — Placement of high-flow tunneled catheter for hemodialysis

SUMMARY:
The patient population for this study is individuals requiring high-flow polyurethane tunneled dialysis catheters (TDC) for hemodialysis access. The primary objective of this study is to compare outcomes of participants who undergo left internal jugular placement of a split-tip versus a step-tip versus symmetric tip catheter. This study will review and compare the complication rate and function of the three catheter designs.

DETAILED DESCRIPTION:
The patient population for this study is individuals requiring high-flow polyurethane tunneled dialysis catheters (TDC) for hemodialysis access. The primary objective of this study is to compare outcomes of participants who undergo left internal jugular placement of a split-tip versus a step-tip versus symmetric tip catheter. Participants will be randomized to receive a split-tip, step-tip or symmetric tip catheter in a 1:1:1 ratio. All participants will be followed per their referring physician's standard of care. Information regarding any patient complications will be obtained from Dr. Allon's dialysis patient database (Vascular Access in Hemodialysis Patients, IRB # X980813005). This study will review and compare the complication rate and function of the three catheter designs. There are no studies to our knowledge that compared catheter designs placed specifically via the left internal jugular vein. The investigators hypothesize that because the left internal jugular vein is anatomically more complex than the right one, tunneled dialysis catheters with split-tip design may perform sub-optimally, compared to step-tip and symmetric tip designs, when placed via the left internal jugular vein. If this hypothesis is true, the results of the study may influence future clinical practice and reduce the rates of replacement of catheters placed through the left internal jugular vein, resulting in better patient care and significant cost-savings.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide a written informed consent
2. 19 years or older
3. Hemodialysis patient needing high-flow polyurethane tunneled dialysis catheter placement via the left internal jugular vein.
4. Patent left internal jugular vein.
5. Able to read and understand English.

Exclusion Criteria:

1. Previous enrollment in this trial
2. Patients unable or unwilling to provide informed consent
3. Prisoners or incarcerated individuals
4. Women who are pregnant
5. Patients in whom the left internal jugular vein is occluded or catheter placement is otherwise contraindicated

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Complication rate | 1 month
  1 month complication rate of left internal jugular vein dialysis catheters

SECONDARY OUTCOMES:
Catheter dysfunction | 1 months
  1 month complication rate of left internal jugular vein dialysis catheters
Catheter dysfunction | 3 months
  3 months complication rate of left internal jugular vein dialysis catheters
Catheter dysfunction | 6 months
  6 months complication rate of left internal jugular vein dialysis catheters
Complication rate | 3 months
  3 months complication rate of left internal jugular vein dialysis catheters
Complication rate | 6 months
  6 months complication rate of left internal jugular vein dialysis catheters

CONTACTS AND LOCATIONS:
Locations (1):
- University of Akabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No